CLINICAL TRIAL: NCT05090280
Title: A Single Dose Study to Evaluate the Pharmacokinetics of Oxycodone and PF614 When PF614 Solution is Co-Administered with Nafamostat, As an Immediate Release Solution And/or Extended Release (ER) Capsule Formulations in Healthy Subjects
Brief Title: Pharmacokinetics of Oxycodone and PF614 Co-Administered with Nafamostat (PF614-MPAR-101)
Acronym: MPAR-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: Quotient Sciences (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QSC203698; 5UH3DA047682-04 (NIH)
Record Dates: First submitted 2021-09-28; First posted 2021-10-22 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Naltrexone; nafamostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF614 solution (Experimental): Cohort 1 and 6 will consist of 6 evaluable subjects. Subjects will receive the PF614 solution alone and concomitantly with nafamostat as an IR solution and/or ER prototype capsules. Subjects will receive naltrexone prior to and following each regimen.
  Cohorts 2 to 5 and Cohorts 7 to 10 will consist of 5 evaluable subjects in each cohort.
  Only 2 sentinel subjects will be dosed (one male and one female) in Period 2, Cohort 1. After review of the PK data and safety data, the safety advisory committee will decide the nafamostat dose level.
  After Cohorts 3 and 8 only: The fed vs fasted regimen will be determined for Cohorts 4 and 9.
  Interventions: Drug: PF614 solution; Drug: Naltrexone Hydrochloride
- PF614 solution concomitantly with nafamostat (Experimental): Cohort 1 and 6 will consist of 6 evaluable subjects. Subjects will receive the PF614 solution alone and concomitantly with nafamostat as an IR solution and/or ER prototype capsules. Subjects will receive naltrexone prior to and following each regimen.
  Cohorts 2 to 5 and Cohorts 7 to 10 will consist of 5 evaluable subjects in each cohort.
  Only 2 sentinel subjects will be dosed (one male and one female) in Period 2, Cohort 1. After review of the PK data and safety data, the safety advisory committee will decide the nafamostat dose level.
  After Cohorts 3 and 8 only: The fed vs fasted regimen will be determined for Cohorts 4 and 9.
  Interventions: Drug: PF614 solution; Drug: Naltrexone Hydrochloride; Drug: Nafamostat Mesylate

INTERVENTIONS:
Drug: PF614 solution — PF614 solution is an oxycodone prodrug
  Other Names: PRF06104; Oxycodone prodrug
Drug: Naltrexone Hydrochloride — Naltrexone 50 mg has been selected to be administered on Day -1 (single dose), Day 1 (BID), and Day 2 (single-dose) to reduce opioid-related adverse effects.
  Other Names: ReVia
Drug: Nafamostat Mesylate — Maximum dose of 10 mg nafamostat co-administered with PF614 solution. Nafamostat will be dosed as an immediate-release (IR) solution or as prototype extended-release (ER) capsules.
  Other Names: Futhan
  Arms: PF614 solution concomitantly with nafamostat

SUMMARY:
A single dose study to assess the pharmacokinetics (PK) of oxycodone, when PF614 is solution is administered alone and with nafamostat as an immediate-release (IR) solution and/or extended-release (ER) capsule prototypes.

DETAILED DESCRIPTION:
This is a single center, randomized, open-label formulation development study for the nafamostat formulation (IR solution and/or ER prototype capsules) and will have the option to assess the effect of food on a selected formulation of healthy subjects. Parts 1 and 2 are planned to enroll a total of 64 healthy subjects, with roughly equal number of males and an even number of females with roughly equal number of males and females in each cohort if possible. Subjects will be randomized to regimen stratified by gender prior to first dose. Cohort 1 and Cohort 6 will consist of 8 subjects who will receive dosing on two occasions in a 2-period sequential design. Cohorts 2 to 5 and Cohorts 7 to 10 will consist of 6 subjects in each cohort and they will receive dosing on a single occasion only. Cohorts 2 to 5 and Cohorts 7 to 10 can be dosed in parallel after Cohort 1 dosing.

Part 1 (with naltrexone blockade) and Part 2 (without naltrexone), Cohorts 1-10, were later expanded to include 6-13 subjects each.

In Cohort 1 and Cohort 6, subjects will receive the PF614 solution alone and concomitantly with nafamostat. In addition, prior to and following each regimen in all periods, subjects will receive blocking doses of the opiate antagonist naltrexone to reduce the opioid-related side effects.

Interim reviews of the safety and PK data for oxycodone and PF614 to 48h post-dose will take place after Cohorts 1 and 6, Cohorts 2 and 7, Cohorts 3 and 8 and Cohorts 4 and 9 to decide upon the following: nafamostat formulation to dose in the subsequent period; After Cohorts 3 and 8 only: The prandial status (fed vs fasted) for Cohort 4 and Cohort 9.

Extended-release prototype capsule formulations will be selected from a 2-dimensional design space describing formulation variables for release rate and dose; however the maximum nafamostat dose to be administered with be 10 mg.

Part 3 (N=12 subjects) was added as a 7-period open-label cross-over study to assess the selected combination of nafamostat IR solution and/or ER prototype capsule(s) identified from Part 2 who were administered with PF614 solution at increasing dose levels to simulate overdose. All subjects in Part 3 received naltrexone blockade.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Ages 18 to 55 years, inclusive, at time of signing informed consent
3. Body mass index of 18.0 to 32.0 kg/m2 as measured at screening or, if outside the range, considered not clinically significant by the investigator
4. Minimum weight of 50kg at screening
5. Must be willing and able to comply with all study requirements
6. Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures
7. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Subjects who have received any Investigational Medical Product (IMP) in a clinical research study within 5 half-lives or within 30 days prior to first dose
2. Subjects who are, or are immediate family members of, a study site or sponsor employee
3. Evidence of current SARS-CoV-2 infection
4. Subjects who have previously been administered IMP in this study
5. History of any drug or alcohol abuse in the past 2 years
6. Regular alcohol consumption in males >21 units per week and females >14 units per week
7. A confirmed positive alcohol urine test at screening or admission
8. Current smokers and those who have smoked within the last 12 months. A confirmed positive urine cotinine test at screening or first admission
9. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
10. Females of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at each admission
11. Females who are expected to have their menses during the dosing period
12. Male subjects with pregnant or lactating partners
13. Have poor venous access that limits phlebotomy
14. Clinically significant abnormal chemistry, hematology, coagulation, or urinalysis as judged by the investigator
15. Positive drugs of abuse test result
16. Positive hepatis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus antibody results
17. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or GI disease, neurological or psychiatric disorder, as judged by the investigator
18. Subjects with a history of cholecystectomy or gall stones
19. Subjects with a history of seizures
20. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
21. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
22. Donation of blood within 2 months or donation of plasma within 7 days prior to first dose of study medication -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Tmax [Time to Maximum Plasma Concentration] | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Time to maximum observed concentrations of oxycodone following administration of PF614 solution alone and with nafamostat
Pharmacokinetic Cmax [Maximum Plasma Concentration] | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Maximum (peak) observed concentration of oxycodone following administration of PF614 solution alone and with nafamostat
Pharmacokinetic C24 [Plasma concentration at 24 hours] | 24 hours
  Concentration of oxycodone at 24h post-dose following administration of PF614 solution alone and with nafamostat
Pharmacokinetic AUC [Area Under the Curve] | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Area under the concentration-time curve from time 0 to the time of last measurable concentrations of oxycodone following administration of PF614 solution alone and with nafamostat
Pharmacokinetic AUC(0-last) | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Area under the concentration-time curve from time 0 extrapolated to time-infinity of oxycodone following administration of PF614 solution alone and with nafamostat
Pharmacokinetic T1/2 [Half-life] | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Terminal elimination half-life concentrations of oxycodone following administration of PF614 solution alone and with nafamostat

SECONDARY OUTCOMES:
Bioavailability Cmax | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Comparative evaluation of the bioavailability of oxycodone and PF614 based on Cmax when PF614 solution is co-administered with nafamostat in the fed state compared to the fasted state
Bioavailability AUC(0-last) | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Comparative evaluation of the bioavailability of oxycodone and PF614 based on AUC(0-last) when PF614 solution is co-administered with nafamostat in the fed state compared to the fasted state
Bioavailability AUC(0-inf) | pre-dose, 0.5,1,1.5,2,3,4,6,8,12,16,24,36,48 hours
  Comparative evaluation of the bioavailability of oxycodone and PF614 based on AUC(0-inf) when PF614 solution is co-administered with nafamostat in the fed state compared to the fasted state
Incidence of Treatment-Emergent Adverse Effects [Safety and Tolerability] | 30 days
  Adverse events (AEs), Significant Adverse Events (SAEs), AEs leading to discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Levy, MD, PhD, Principal Investigator — Medical Director, Quotient Sciences
Locations (1):
- Quotient Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523
- [Background] Kirkpatrick DL, Schmidt WK, Morales R, Cremin J, Seroogy J, Husfeld C, Jenkins T. In vitro and in vivo assessment of the abuse potential of PF614, a novel BIO-MD prodrug of oxycodone. J Opioid Manag. 2017 Jan/Feb;13(1):39-49. doi: 10.5055/jom.2017.0366. PMID 28345745